CLINICAL TRIAL: NCT00455988
Title: Developement of Questionnaire to Evaluate a Regularity of Lifestyle in Type 2 Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eulji University Hospital (Other)
Other Study IDs: Questionnaire06-27-1
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Type 2 Diabetes
Keywords: questionnaire developement; regularity; lifestyle; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
In order to manage of type 2 diabetic patients with irregular lifestyle, developement of an appropriate questionnaire to evaluate a regularity of lifestyle is necessary.

DETAILED DESCRIPTION:
We have a plan to perform the seven day's records and the questionnaires which is necessary to type 2 diabetic patients for the initial step. Next, we will revise a questionnaire with professional advices for several times. Finally we will test a reliability with a final version as form of multisite based study and will confirm a questionnaire for a regularity of lifestyle in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients

Exclusion Criteria:

* Type 1 diabetic patients, gestational DM patients

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2006-09; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Wan Min, MD., PhD, Principal Investigator — Eulji University Hospital Diabetes Center
Locations (1):
- Eulji University Hospital, Seoul, South Korea